CLINICAL TRIAL: NCT03517540
Title: A Randomized, Double-blind, Multicenter Study to Assess the Safety, Tolerability, and Efficacy of a Combination Treatment of Tropifexor (LJN452) and Cenicriviroc (CVC) in Adult Patients With Nonalcoholic Steatohepatitis (NASH) and Liver Fibrosis
Brief Title: Study of Safety, Tolerability, and Efficacy of a Combination Treatment of LJN452 and CVC in Adult Patients With NASH and Liver Fibrosis
Acronym: TANDEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLJC242A2201J; 2017-004208-24 (EudraCT Number); LJC242A2201J (Other: Novartis)
Record Dates: First submitted 2018-04-09; First posted 2018-05-07 (Actual); Results first posted 2021-11-12 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: Steatohepatitis; NASH; NAFLD; Fatty Liver Disease; Liver; Liver fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis | interventions — tropifexor; cenicriviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Tropifexor (LJN452) - Dose 1 (Experimental): tropifexor 140 mcg, once daily; given orally
  Interventions: Drug: Tropifexor (LJN452)
- Arm B: Cenicriviroc (CVC) (Experimental): CVC 150 mg, once daily; given orally
  Interventions: Drug: Cenicriviroc (CVC)
- Arm C: Tropifexor (LJN452) Dose 1 + CVC (Experimental): tropifexor 140 mcg + CVC 150 mg, once daily; given orally
  Interventions: Drug: Tropifexor (LJN452); Drug: Cenicriviroc (CVC)
- Arm D: Tropifexor Dose 2 + CVC (Experimental): tropifexor 90 mcg + CVC 150 mg, once daily; given orally
  Interventions: Drug: Tropifexor (LJN452); Drug: Cenicriviroc (CVC)

INTERVENTIONS:
Drug: Tropifexor (LJN452) — Comparison with monotherapy and different combination doses
  Other Names: LJN452
  Arms: Arm A: Tropifexor (LJN452) - Dose 1; Arm C: Tropifexor (LJN452) Dose 1 + CVC; Arm D: Tropifexor Dose 2 + CVC
Drug: Cenicriviroc (CVC) — Comparison with monotherapy and different combination doses
  Other Names: CVC
  Arms: Arm B: Cenicriviroc (CVC); Arm C: Tropifexor (LJN452) Dose 1 + CVC; Arm D: Tropifexor Dose 2 + CVC

SUMMARY:
The purpose of this study was to assess the safety, tolerability, and efficacy of a combination treatment of tropifexor (LJN452) and cenicriviroc (CVC) in adult patients with nonalcoholic steatohepatitis (NASH) and liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent Male and female patients 18 years or older (at the time of the screening visit). Patients must weigh at least 50 kg (110 lb) and no more than 200 kg (440 lb) to participate in the study.

Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Adequate liver biopsy sample for evaluation by Central Reader. Presence of NASH as demonstrated by histologic evidence based on liver biopsy - NASH with fibrosis stage F2/F3, demonstrated on liver biopsy during the screening period. Alternatively, a historical biopsy can be used if performed within 6 months prior to screening.

Exclusion Criteria:

Use of other investigational drugs within 5 half-lives of enrollment or within 30 days whichever is longer.

History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes.

Previous exposure to elafibranor, CVC, tropifexor, obeticholic acid (OCA), LMB763 or other FXR agonist.

Participated in a clinical trial and treated with any investigational product being evaluated for the treatment of liver fibrosis or NASH in the 6 months before screening.

Patients taking medications prohibited by the protocol. History of treated or untreated malignancy of any organ system, other than localized basal cell carcinoma of the skin or treated cervical intraepithelial neoplasia, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases .

Pregnant or nursing (lactating) women. Women of child-bearing potential. Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening (significant alcohol consumption is defined as more than 20 g/day in females and more than 30 g/day in males, on average) and/or a score on the modified AUDIT questionnaire ≥ 8.

Inability to reliably quantify alcohol consumption. History or evidence of ongoing drug abuse, within the last 6 months prior to randomization.

Prior or planned (during the study) bariatric surgery. Uncontrolled diabetes defined as HbA1c ≥ 9% at screening Clinical evidence of hepatic decompensation or severe liver impairment. Previous diagnosis of other forms of chronic liver disease. Calculated eGFR less than 60 mL/min (using the MDRD formula). History of biliary diversion History of liver transplantation or planned liver transplant. Known positivity for HIV. History or current diagnosis of ECG abnormalities indicating significant risk of safety for the patient to participate.

History of inflammatory bowel disease. Patients who are not candidates for liver biopsy. Presence of cirrhosis on liver biopsy (F4 by NASH CRN System) or medical history Patients with an abnormal platelet count (referring to reference ranges from the central lab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- United States (24):
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, North Little Rock, Arkansas
  - Novartis Investigative Site, Coronado, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Rialto, California
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Concord, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Morehead City, North Carolina
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Chattanooga, Tennessee
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Hermitage, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Seattle, Washington
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, San Juan Bautista, Buenos Aires
- Belgium (2):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Leuven
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Shebeen El-Kom, Egypt
- France (3):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Strasbourg
- Germany (2):
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, New Delhi, National Capital Territory of Delhi, India
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (5):
  - Novartis Investigative Site, Modena, Itlay
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Milan
- Novartis Investigative Site, Riga, Latvia
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Izmir
- United Kingdom (3):
  - Novartis Investigative Site, High Heaton, Newcastle Upon Tyne
  - Novartis Investigative Site, Aberdeen
  - Novartis Investigative Site, Torquay

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Pedrosa M, Seyedkazemi S, Francque S, Sanyal A, Rinella M, Charlton M, Loomba R, Ratziu V, Kochuparampil J, Fischer L, Vaidyanathan S, Anstee QM. A randomized, double-blind, multicenter, phase 2b study to evaluate the safety and efficacy of a combination of tropifexor and cenicriviroc in patients with nonalcoholic steatohepatitis and liver fibrosis: Study design of the TANDEM trial. Contemp Clin Trials. 2020 Jan;88:105889. doi: 10.1016/j.cct.2019.105889. Epub 2019 Nov 13. PMID 31731005
- [Derived] Parthasarathy G, Malhi H. Macrophage Heterogeneity in NASH: More Than Just Nomenclature. Hepatology. 2021 Jul;74(1):515-518. doi: 10.1002/hep.31790. Epub 2021 May 22. No abstract available. PMID 33666272
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=984

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 193 participants enrolled at 65 sites in 17 countries
Pre-assignment Details: 450 of 643 subjects discontinued during screening phase
Groups:
- Arm A: Tropifexor (LJN452) - Dose 1: tropifexor 140 mg, once daily
- Arm B: Cenicriviroc (CVC): CVC 150 mg, once daily
- Arm C: Tropifexor (LJN452) Dose 1 + CVC: tropifexor 140 mg + CVC 150 mg, once daily
- Arm D: Tropifexor Dose 2 + CVC: tropifexor 90 mg + CVC 150 mg, once daily
Period: Overall Study
Arm/Group | Arm A: Tropifexor (LJN452) - Dose 1 | Arm B: Cenicriviroc (CVC) | Arm C: Tropifexor (LJN452) Dose 1 + CVC | Arm D: Tropifexor Dose 2 + CVC
Started | 50 | 48 | 47 | 48
Completed | 36 | 41 | 38 | 43
Not Completed | 14 | 7 | 9 | 5
Not completed — Protocol Violation | 2 | 0 | 0 | 1
Not completed — Adverse Event | 9 | 3 | 8 | 1
Not completed — Withdrawal by Subject | 3 | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) - All participants to whom study treatment was assigned (excluding patients who were mis-randomized and did not take investigational drug. Mis-randomized participants were those who were not qualified for randomization but were inadvertently randomized into the study). Following the intent-to-treat (ITT) principle, patients were analyzed according to the treatment they had been assigned to at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Tropifexor (LJN452) - Dose 1 | Arm B: Cenicriviroc (CVC) | Arm C: Tropifexor (LJN452) Dose 1 + CVC | Arm D: Tropifexor Dose 2 + CVC | Total
Number analyzed (Participants) | 50 | 48 | 47 | 48 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (13.35) | 53.7 (11.79) | 54.7 (12.65) | 54.9 (12.29) | 54.5 (12.52)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 35 | 39 | 37 | 38 | 149
  >=65 | 15 | 9 | 10 | 10 | 44
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 20 | 17 | 18 | 25 | 80
  Female | 30 | 31 | 29 | 23 | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 41 | 44 | 40 | 43 | 168
  Asian | 7 | 4 | 5 | 5 | 21
  Black | 1 | 0 | 2 | 0 | 3
  Unknown | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Occurrence of adverse events and serious adverse events
  Adverse Events (AEs) are any untoward sign or symptom that occurs during the study treatment and then up to 66 weeks
Time Frame: AEs were collected from first dose of study treatment until end of study treatment at week 48 and then up to maximum duration of 66 weeks
Population: Safety set (SAF) - All patients who received at least one dose of study drug and had at least one post-baseline safety assessment. Of note, the statement that a patient had no AEs also constituted a safety assessment. Patients were analyzed according to the treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tropifexor (LJN452) - Dose 1 | Arm B: Cenicriviroc (CVC) | Arm C: Tropifexor (LJN452) Dose 1 + CVC | Arm D: Tropifexor Dose 2 + CVC
Number analyzed (Participants) | 50 | 48 | 47 | 48
Participants
  Number of participants with at least one Adverse Event (AE) | 42 | 41 | 40 | 42
  Number of participants with at least one Serious Adverse Events (SAEs) | 5 | 3 | 4 | 10
  Deaths | 0 | 0 | 0 | 0

2. Secondary Outcome: Proportion of Participants Who Have at Least a One Point Improvement in Fibrosis
Description: Efficacy of tropifexor + CVC in patients with Nonalcoholic steatohepatitis (NASH) with fibrosis stage F2/F3 as assessed by histological improvement after 48 weeks of treatment compared to monotherapies (tropifexor and CVC) compared to baseline biopsy
Time Frame: baseline to 48 Weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tropifexor (LJN452) - Dose 1 | Arm B: Cenicriviroc (CVC) | Arm C: Tropifexor (LJN452) Dose 1 + CVC | Arm D: Tropifexor Dose 2 + CVC
Number analyzed (Participants) | 31 | 38 | 37 | 40
Participants | 10 | 12 | 11 | 13
Statistical Analysis 1: Comparison: Arm A: Tropifexor (LJN452) - Dose 1 vs Arm C: Tropifexor (LJN452) Dose 1 + CVC; Test type: Superiority; p = 0.688, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.25 to 2.63]
Statistical Analysis 2: Comparison: Arm A: Tropifexor (LJN452) - Dose 1 vs Arm D: Tropifexor Dose 2 + CVC; Test type: Superiority; p = 0.985, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.51 to 1.99]
Statistical Analysis 3: Comparison: Arm C: Tropifexor (LJN452) Dose 1 + CVC vs Arm D: Tropifexor Dose 2 + CVC; Test type: Superiority; p = 0.870, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.3 to 2.84]
Statistical Analysis 4: Comparison: Arm B: Cenicriviroc (CVC) vs Arm D: Tropifexor Dose 2 + CVC; Test type: Superiority; p = 0.710, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.41 to 3.61]

3. Secondary Outcome: Proportion of Participants With Resolution of Steatohepatitis
Description: as for outcome 2
Time Frame: baseline to 48 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tropifexor (LJN452) - Dose 1 | Arm B: Cenicriviroc (CVC) | Arm C: Tropifexor (LJN452) Dose 1 + CVC | Arm D: Tropifexor Dose 2 + CVC
Number analyzed (Participants) | 31 | 38 | 37 | 40
Participants | 8 | 8 | 5 | 9
Statistical Analysis 1: Comparison: Arm A: Tropifexor (LJN452) - Dose 1 vs Arm C: Tropifexor (LJN452) Dose 1 + CVC; Test type: Superiority; p = 0.136, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.08 to 1.61]
Statistical Analysis 2: Comparison: Arm A: Tropifexor (LJN452) - Dose 1 vs Arm D: Tropifexor Dose 2 + CVC; Test type: Superiority; p = 0.747, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.24 to 2.9]
Statistical Analysis 3: Comparison: Arm B: Cenicriviroc (CVC) vs Arm C: Tropifexor (LJN452) Dose 1 + CVC; Test type: Superiority; p = 0.784, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.18 to 3.63]
Statistical Analysis 4: Comparison: Arm B: Cenicriviroc (CVC) vs Arm D: Tropifexor Dose 2 + CVC; Test type: Superiority; p = 0.521, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.4 to 5.69]

ADVERSE EVENTS:
Time Frame: AEs were collected from first dose of study treatment until end of study treatment at week 48 and then up to maximum duration of 66 weeks
Description: Adverse Events (AEs) are any untoward sign or symptom that occurs during the study treatment and up to of 66 weeks
Groups:
- Tropifexor 140mg: Tropifexor 140mg
- CVC 150mg: CVC 150mg
- Tropifexor 140mcg + CVC 150mg: Tropifexor 140mg + CVC 150mg
- Tropifexor 90 mg + CVC 150 mg: Tropifexor 90 mg + CVC 150 mg
Arm/Group | Tropifexor 140mg | CVC 150mg | Tropifexor 140mcg + CVC 150mg | Tropifexor 90 mg + CVC 150 mg
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/48 | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 5/50 | 3/48 | 4/47 | 10/48
Other Adverse Events (participants affected / at risk) | 39/50 | 30/48 | 33/47 | 32/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tropifexor 140mg (N=50) | CVC 150mg (N=48) | Tropifexor 140mcg + CVC 150mg (N=47) | Tropifexor 90 mg + CVC 150 mg (N=48)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tropifexor 140mg (N=50) | CVC 150mg (N=48) | Tropifexor 140mcg + CVC 150mg (N=47) | Tropifexor 90 mg + CVC 150 mg (N=48)
Cataract (Eye disorders) | 0 | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 5 | 2
Constipation (Gastrointestinal disorders) | 5 | 2 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 7 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 3 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 6 | 7 | 6
Asthenia (General disorders) | 4 | 2 | 5 | 3
Fatigue (General disorders) | 7 | 4 | 5 | 4
Oedema peripheral (General disorders) | 0 | 0 | 0 | 4
Bronchitis (Infections and infestations) | 1 | 0 | 3 | 1
Ear infection (Infections and infestations) | 0 | 0 | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 3 | 3
Nasopharyngitis (Infections and infestations) | 2 | 3 | 2 | 2
Sinusitis (Infections and infestations) | 2 | 1 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 5 | 5
Urinary tract infection (Infections and infestations) | 7 | 3 | 2 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 10 | 15 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT03517540/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03517540/SAP_001.pdf